CLINICAL TRIAL: NCT04630288
Title: ANTIPLATELET TREATMENT IN ACUTE CORONARY SYNDROMES. SAFETY AND EFFICACY OF ANTIPLATELET SWITCHING Safety and Efficacy of Ticagrelor vs Clopidogrel in Patients With Acute Coronary Syndrome
Brief Title: Safety and Efficacy of Ticagrelor vs Clopidogrel in Patients With Acute Coronary Syndrome
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Andalusian Initiative for Advanced Therapies - Fundación Pública Andaluza Progreso y Salud (Other)
Responsible Party: Sponsor
Organization: Andalusian Network for Design and Translation of Advanced Therapies (Other)
Other Study IDs: FPS-AAS-2019-01 (ESR-17-13127)
Record Dates: First submitted 2020-01-14; First posted 2020-11-16 (Actual); Last update posted 2020-11-16 (Actual); Status verified 2020-11

CONDITIONS: Acute Coronary Syndromes
MeSH Terms: conditions — Acute Coronary Syndrome | interventions — Clopidogrel; Ticagrelor

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Clopidogrel: Clopidogrel is a prodrug that requires metabolic activation in two stepsby hepatic CYP450 enzymes to produce the active metabolite that inhibits platelet aggregation. The active metabolite of clopidogrel selectively inhibits the binding of adenosine diphosphate (ADP) to its platelet P2Y12 receptor and the subsequent ADP-mediated activation of the glycoprotein GPIIb/IIIa complex, thereby inhibiting platelet aggregation. Consequently, due to the irreversible binding to the P2Y12 receptor,platelets exposed to clopidogrel's active metabolite are affected for the remainder of their lifespan (about 7 to 10 days) and recovery of normal platelet function occurs at a rate consistent with the normal platelet turnover. Clopidogrel was approved by the European Commission on 15 July 1998 for the secondary prevention of atherothrombotic events in adult patients with ACS.
  Interventions: Drug: Clopidogrel
- Ticagrelor: Ticagrelor is a nucleoside analogue member of the chemical class cyclopentyltriazolopyrimidines (CPTP), which is a selective and reversible ADP- receptor antagonist acting on the platelet P2Y12 receptor. This prevents the binding of ADP to the receptor which attenuates plateletactivation and aggregation.The drug was approved by the European Commission on December 3, 2010, for the prevention of thrombotic events (cardiovascular death, myocardial infarction and stroke) in patients with ACS (unstable angina, non ST elevation Myocardial Infarction [NSTEMI] or ST elevation Myocardial Infarction [STEMI]) including patients managed medically, and those who are managed with percutaneous coronary intervention (PCI) or coronary artery by-pass grafting (CABG).
  Interventions: Drug: Ticagrelor

INTERVENTIONS:
Drug: Clopidogrel — Describe the safety of Ticagrelor vs Clopidogrel use, in patients with ACS in terms of major bleeding between 30 days and one year after the index ACS event. An ITT approach and IPCW method to adjust for change of initial treatment will be used for the analysis.
  Groups: Clopidogrel
Drug: Ticagrelor — Describe the safety of Ticagrelor vs Clopidogrel use, in patients with ACS in terms of major bleeding between 30 days and one year after the index ACS event. An ITT approach and IPCW method to adjust for change of initial treatment will be used for the analysis.
  Groups: Ticagrelor

SUMMARY:
Multicenter post-approval observational retrospective cohort study in routine clinical practice (Real World Evidence Study) to assess the 1-year safety profile associated with ticagrelor and clopidogrel therapy in a contemporary reprospective cohort of patients who survived the initial 30-day period after the index hospitalization for acute coronary syndrome (ACS).

DETAILED DESCRIPTION:
To date, there are still a paucity of data on the medium- and long-term safety and efficacy outcomes of new antiplatelet agents, namely Ticagrelor and Prasugrel, compared to Clopidogrel in a real-world ACS setting.

The ARIAM-Andalusia multicentre Registry, and the CREA-ARIAM multicentre Registry (ClinicalTrials.gov Identifier: NCT02500290; Fundación Pública Andaluza Progreso y SaludIdentifier: FPS-AAS-2014-01), are two Real World Evidence (RWE) studies aimed to investigate real-world practice on antiplatelet treatment in patients with ACS in Andalusia (Western Spain).

Our group are interested in performing a retrospective observational pilot analysis using data from patients with ACS admitted to cardiovascular intensive care units in Andalusia (Spain), who were prospectively included in the ARIAM-Andalusia multicentre Registry, and the CREA-ARIAM multicentre Registry (ClinicalTrials.gov Identifier: NCT02500290; Fundación Pública Andaluza Progreso y Salud-Identifier: FPS-AAS-2014-01) between 2014 and March 2019. The main findings from the RWE study revealed a consistent net clinical benefit of Ticagrelor vs Clopidogrel resulted in a significant reduction of short-term all-cause mortality favored Ticagrelor. In this scenario, after baseline imbalance adjustment using propensity score matching (PSM) and IPTW (inverse probability of treatment weight) methods, the net clinical benefit with Ticagrelor persisted. Preliminary results of the above mentioned study have been presented as an oral communication at the Annual Scientific Meeting of the Spanish Society of Cardiology (Madrid, October 2017).

The aim of this new pilot study suggested is to describe the efficacy and safety of Ticagrelor vs Clopidogrel after the first 30 days from hospital discharge and up to 1 year follow-up.

ELIGIBILITY:
Inclusion Criteria:

All-comers ACS population (with or without ST segment elevation, including unstable angina) with:

A recent CCU admission (patients included in the ARIAM-CREA study within 1 week from the index ACS admission between March 1, 2015 to March 31, 2018), irrespective of either the initial management (invasive or non-invasive) or the revascularization procedure (PCI with stenting or CABG) discharged on DAPT including either Ticagrelor or Clopidogrel and have survived the first 30-day follow-up period from the index ACS event and could complete a 12-month follow-up.

Exclusion Criteria:

* Age < 18 years.
* Subjects who died in the first 30-day follow-up period from the index ACS event, including those who died during the index admission.
* A medical condition likely to limit survival to less than 1 year.
* Any factors judged by the local investigators to be likely to limit adherence to pharmacological treatment.
* Failure to obtain informed consent from participant.
* Currently enrolled in an interventional clinical research trial involving an investigational product (drug) or device
* Not available for follow-up over a minimum of 365 days, e.g. no fixed home address.
* Pregnancy, breast-feeding, or intend to become pregnant during the study period population should be always considered as exclusion criterion.
* Non-ACS diagnosis at discharge, i.e., acute myocarditis, Takotsubo syndrome, pulmonary thromboembolism or acute aortic syndromes.
* Myocardial infarction secondary to an ischaemic imbalance or type 2 myocardial infarction (Third Universal Definition of MI), in instances of myocardial injury with necrosis, where a condition other than CAD contributes to an imbalance between myocardial oxygen supply and/or demand, i.e., anaemia, sepsis, tachyarrhythmias, hypotension, heart failure…
* Patients not discharged on dual antiplatelet therapy (DAPT) consistent on low dose of ASA plus a P2Y12platelet receptor inhibitor (Clopidogrel or Ticagrelor)
* Patient discharged on DAPT including Prasugrel as the P2Y12 inhibitor drug.
* Hypersensitivity to ticagrelor or any of the excipients.
* Active pathological bleeding.
* History of intracranial haemorrhage (ICH).
* Severe hepatic impairment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with ACS in a real world setting
Sampling Method: Non-Probability Sample
Enrollment: 1900 (Actual)
Dates: Start 2019-07-02 (Actual); Primary Completion 2019-11-01 (Actual); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Major bleeding | During 2 months
  Defined as BARC type≥ 3 according to the Bleeding Academic Research Consortium (BARC) definition at 1-year follow-up after the index ACS.

SECONDARY OUTCOMES:
Thrombolysis in Myocardial Infarction (TIMI) | During 2 months
  Bleeding criteria
BARC definition | During 2 months
  Bleeding criteria
Major Adverse Cardiac and Cerebrovascular Events (MACCE) | During 2 months
  Defined as the composite of all-cause mortality, myocardial infarction (MI), target lesion revascularization (TLR), stent thrombosis and stroke or TIA at 1-year follow-up after the index ACS admission.
All-cause mortality | During 2 months
  Component of MACCE
Myocardial infarction | During 2 months
  Component of MACCE
Target lesion revascularization | During 2 months
  Component of MACCE
Stent thrombosis | During 2 months
  Component of MACCE
Stroke | During 2 months
  Component of MACCE
Net clinical benefit/Net Adverse Clinical Event (NACE): | During 2 months
  Defined as the composite of the efficacy (Major Adverse Cardiac and Cerebrovascular Events-MACCE) and safety (BARC type≥ 2 bleeding episodes according to the Bleeding Academic Research Consortium (BARC) definition for bleeding) outcomes at 1 year after the index ACS.

CONTACTS AND LOCATIONS:
Locations (2):
- Spain (2):
  - Fundación Pública Progreso y Salud, Seville
  - Hospital Universitario Virgen Macarena, Seville

REFERENCES:
- [Derived] Almendro-Delia M, Blanco-Ponce E, Carmona-Carmona J, Arboleda Sanchez JA, Rodriguez Yanez JC, Soto Blanco JM, Fernandez Garcia I, Castillo Caballero JM, Garcia-Rubira JC, Hidalgo-Urbano RJ. Comparative Safety and Effectiveness of Ticagrelor versus Clopidogrel in Patients With Acute Coronary Syndrome: An On-Treatment Analysis From a Multicenter Registry. Front Cardiovasc Med. 2022 May 27;9:887748. doi: 10.3389/fcvm.2022.887748. eCollection 2022. PMID 35711382